CLINICAL TRIAL: NCT06719427
Title: Quantitative Electroencephalography to Longitudinally Assess the Functional Brain Signature of Treatment-resistant Depression and Recovery With Therapeutic Neuromodulation
Brief Title: qEEG Brain Signature of Depression & Neuromodulation-induced Recovery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Mitacs (Industry); iMediSync (Unknown)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6178; IT41597 (Other Grant/Funding Number: Mitacs)
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Diorder
Keywords: Transcranial Magnetic Stimulation; Treatment-resistant Depression; Mood Disorders; Mental Disorders; Depressive Disorder; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; qEEG; resting-state connectivity; neuromodulation; brain networks
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Mood Disorders; Mental Disorders; Depressive Disorder; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cluster Maintenance TMS (Active Comparator): Participants will receive a cluster of treatments consisting of 5 treatments over two consecutive week days (either 2 treatments on day 1 followed by 3 treatments day 2 or vice-versa, based on scheduling)
  Interventions: Device: Transcranial Magnetic Stimulation
- Gradual Tapering TMS (Active Comparator): Participants will receive a once daily treatment protocol delivered once weekly for 1 month, and gradually tapering the frequency of treatment to 1 treatment every 2 weeks for 2 months
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — rTMS is a non-invasive brain stimulation that uses magnetic fields to stimulate specific areas of the brain. It is commonly used for the treatment of neurological and psychiatric disorders, such as major depressive disorder (MDD), anxiety, and sometimes ALS.
  Other Names: rTMS; iTBS

SUMMARY:
This study aims to explore how repetitive transcranial magnetic stimulation (rTMS), a treatment for depression, affects brain function. Depression disrupts the brain's complex network or regions that regulate cognition, emotion, and behavior. rTMS targets these disruptions to restore network function. To measure these effects, researchers will use dry quantitative EEG (qEEG), a new technology that records brain electrical activity quickly (15 minutes compared to 1 hour for traditional EEG) without the need for gel or lengthy electrode setups. This study will evaluate a novel qEEG activity developed by iMediSync (Republic of South Korea) in patients treated with neuromodulation for depression before, during, and up to 12 months after treatment to see if changes in brain activity to identify patterns associated with symptomatic improvement and relapse risk. Findings could help personalize depression treatments by predicting patient outcomes and optimizing care.

DETAILED DESCRIPTION:
The objective of this study is to evaluate functional brain activity measures that correlate with clinically assessed mood symptoms and their changes before, during, and after repetitive transcranial magnetic stimulation (rTMS) treatment for a major depressive episode. A secondary aim is to explore the relationship between pre- and post-treatment functional brain changes and depression outcomes, including changes in depression scores, response rates, and remission status. The dorsolateral prefrontal cortex (DLPFC), a brain region involved in mood regulation, shows altered activity in depression and will be targeted in this study. All patients in this study will undergo an accelerated rTMS protocol over the course of five days, using the pre-treatment imaging to localize the brain region (i.e. DLPFC) targeted by the TMS coil. In addition to rTMS, the investigators will administer questionnaires to evaluate mood and function at multiple time points: before, during, and after treatment. Patients will also undergo dry quantitative EEG (qEEG), which records brain electrical activity to see how these networks are altered in depression and rescued by rTMS. Participants will also undergo dry quantitative EEG (qEEG) recordings, a method that measures brain electrical activity, to investigate how brain networks are disrupted in depression and how they are modulated by rTMS. Participants who respond to rTMS will be monitored for recurrence of depressive symptoms during follow-up visits. If depressive symptoms worsen, maintenance treatment will be administered. Two maintenance TMS protocols will be compared in this study: 1) a gradually tapering protocol involving once-daily treatments delivered weekly for one month, followed by a gradual taper to one treatment every two weeks for two months, 2) a cluster protocol involving five treatments delivered over two consecutive weekdays (e.g., two treatments on Day 1 and three treatments on Day 2, or vice versa). This research aims to deepen our understanding of the mechanisms by which rTMS modulates brain activity, improve our ability to predict treatment response, and determine the most effective maintenance treatment protocol for sustained symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Depression based on Diagnostic and Statistical Manual (DSM) 5.0 criteria.
* Receiving a neuromodulation (rTMS) treatment for depression at the HCN
* Physically healthy
* Age 18-80, inclusive.
* Able to provide informed consent and comply with the study protocol.
* Patients will not be excluded solely based on communication (i.e., non-English speaking) unless they have exclusion criteria that is the cause of the communication difficulties.

Exclusion Criteria:

* Moderate substance use disorder or greater severity based on DSM 5.0 criteria and confirmed by a study MD on clinical assessment.
* Mild and major comorbid medical conditions (as determined by investigators - e.g., neurological diseases, uncontrolled hypertension or diabetes, malignancy)
* A major comorbid psychiatric disorder (as determined by investigators - e.g., schizophrenia or bipolar disorder) and/or psychosis at the time of study enrollment.
* History of seizure disorder
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Score on the Montgomery-Asberg Depression Rating Scale (MADRS) | 2 years
  Change in depression symptomatology as assessed by the clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) (range 0-60). Higher scores indicate worse outcomes

SECONDARY OUTCOMES:
Changes in functional connectivity | 2 years
  Change between baseline measured qEEG resting-state connectivity and post TMS qEEG connectivity
Relapse rates measured on the Montgomery-Asberg Depression Rating Scale | 2 years
  Examine relapse rates on the depression rating scale (0-60) over 12 months, following successful response to neuromodulation with qEEG

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, North York, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No